CLINICAL TRIAL: NCT02400957
Title: Effectiveness of the Addition of Silver Nanoparticles to a Orthodontic Primer in Preventing Enamel Demineralization Adjacent Brackets. ECCA
Brief Title: Addition of Silver Nanoparticles to a Orthodontic Primer in Preventing Enamel Demineralization Adjacent Brackets
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Gabriela Moreno-Meraz, MsC, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEI-FE-023-013
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Tooth Demineralization
Keywords: silver nanoparticles; demineralization; brackets
MeSH Terms: conditions — Tooth Demineralization | interventions — colloidal silver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silver nanoparticles (Experimental): Half of the mouth was applied silver nanoparticles. Allocation was randomized.
  Interventions: Other: Silver nanoparticles
- Placebo (Experimental): Half of the mouth was applied placebo. Allocation was randomized.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Silver nanoparticles — Half of the mouth was applied silver nanoparticles. Allocation was randomized. Evaluate the effectiveness of silver nanoparticles incorporated into the primer orthodontic Transbond XT in preventing enamel demineralization adjacent to brackets.
  Arms: Silver nanoparticles
Other: Placebo — Half of the mouth was applied placebo. Allocation was randomized. Evaluate the effectiveness of silver nanoparticles incorporated into the primer orthodontic Transbond XT in preventing enamel demineralization adjacent to brackets.
  Other Names: Primer-bond
  Arms: Placebo

SUMMARY:
Evaluate the effectiveness of silver nanoparticles incorporated into the primer orthodontic Transbond XT in preventing enamel demineralization adjacent to brackets.

DETAILED DESCRIPTION:
Randomized, split mouth, double-blind, placebo controlled trial. Half of the mouth was applied silver nanoparticles incorporated into the primer orthodontic Transbond XT and the other half with primer-bond as placebo. Evaluate the effectiveness with Diagnodent - pen in preventing enamel demineralization adjacent to brackets.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for orthodontic treatment.

Exclusion Criteria:

* Patients with O.D 11 and / or 21 absent.

  * Patients who present dentures of any kind in OD 11 and 21.
  * Patients presenting endodontic OD 11 and 21.
  * Patients presenting data gingivitis day cementing brackets.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
enamel demineralization (Diagnodent - pen evaluation) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Pierdant, Profesor, Study Director — Universidad Autonoma San Luis Potosi
Locations (1):
- Gabriela Moreno Meraz, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Result] Hernandez-Sierra JF, Galicia-Cruz O, Angelica SA, Ruiz F, Pierdant-Perez M, Pozos-Guillen AJ. In vitro cytotoxicity of silver nanoparticles on human periodontal fibroblasts. J Clin Pediatr Dent. 2011 Fall;36(1):37-41. doi: 10.17796/jcpd.36.1.d677647166398886. PMID 22900442